CLINICAL TRIAL: NCT04491760
Title: Feasibility of Inspiratory Muscle Training in Patients With Acute Myocardial Infarction Undergoing Percutaneous Coronary Intervention and Complicated With High Risk of Pneumonia: a Randomized Controlled Trail
Brief Title: Inspiratory Muscle Training in Patients With Acute Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: No.GDREC2019521H(R1)
Record Dates: First submitted 2020-06-16; First posted 2020-07-29 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2020-06

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training (Experimental): Inspiratory muscle training (IMT) will be perform for 15 minutes each time, twice a day, training every day from 12h to 24h after primary percutaneous coronary intervention (PCI) to 30 days since randomized.
  Interventions: Other: Inspiratory Muscle Training
- Control group (No Intervention): Participants will receive standard care according to the current guideline and clinical practice after primary PCI.

INTERVENTIONS:
Other: Inspiratory Muscle Training — The inspiratory muscle training (IMT) will be carried out with a load of 30% of maximal inspiratory pressure (MIP) using a threshold inspiratory muscle trainer (c-type, Shengchang medical equipment factory, Yuyao city, China) at the beginning. During the hospital period, the resistance will increase incrementally, based on the rate of perceived exertion scored on the Borg scale (Borg, 1982). If the rate of perceived exertion less than 5, the resistance of the inspiratory threshold trainer will then be increase incrementally by 5%. The load for home-based IMT training will be set as the highest training load in the hospital. All patients will be required in sitting position during training, wearing nose-clips.
  Arms: Inspiratory muscle training

SUMMARY:
Pneumonia is uncommon high among patients with acute myocardial infarction (AMI), which increases adverse clinical events and prolongs the hospital stay. Inspiratory muscle training (IMT) is able to improve inspiratory muscle strength and prevent pneumonia in patients undergoing cardiac surgery including coronary artery bypass grafting. Thus, the investigators design the study mainly aim to evaluate the 30 days IMT for the change of inspiratory muscle strength, and also to observe its potentially effect on reducing pneumonia, in participants who accepted primary percutaneous coronary intervention (PCI) and at a high risk of pneumonia.

DETAILED DESCRIPTION:
This is a single center, prospective, randomized controlled study. All participants will be followed up until 30 days after randomized.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years, patients with AMI undergoing primary PCI, admitted to cardiac intensive care unit and at a high pneumonia risk [2 or more of the following parameters are regarded as high risk for pneumonia: 1. Age > 55 years, 2. Diabetes mellitus, 3. Smoking at present, 4. Chronic kidney disease: estimated glomerular filtration rate < 60 mL/min/1.73m2, 5. Forced expiratory volume in the first second of expiration (FEV1) < 80% predicted and FEV1/forced vital capacity (FVC) < 70% predicted]
* be able to understand and agree with informed consent

Exclusion Criteria:

* a history of cerebrovascular accident
* treat with immunosuppressive medication for 30 days before
* neuromuscular disorder
* cardiovascular instability (such as aortic dissection or unstable hemodynamics)
* a history of Coronary Artery Bypass Grafting (CABG)
* expected survival is less than 6 months due to noncardiogenic disease
* participated in other drugs and devices studies within 30 days
* confirmed as ventricular aneurysm
* other conditions not suit for the study after the discussion among the researchers (eg: poor compliance, unable to cooperate for the training)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in inspiratory muscle strength | at baseline, at 30 days
  Static maximal inspiratory pressure (MIP) will be selected for the estimation of inspiratory muscle strength. A standard measurement using Powerbreathe® K5 and according to "ERS Statement on Respiratory Muscle Testing at Rest and during Exercise" published by European Respiratory Society (ERS) will be taken (Laveneziana, 2019). MIP test will be performed at baseline and at 30 days.

SECONDARY OUTCOMES:
Pneumonia | up to 30 days
  The diagnosis of pneumonia is based on guidelines of the American Thoracic Society [American Thoracic Society (ATS) and Infectious Diseases Society of America (IDSA), 2005]. The events of pneumonia will be followed and recorded by experienced doctors when in hospital. After discharged, participants will be followed by the experienced researches, once pneumonia is considered as possible, guidance will be provided for the participants to complete necessary examines, until 30 days.
Major adverse cardiovascular events (MACE) | up to 30 days
  MACE is defined as: all cause death, recurrence of myocardial infarction, stroke at 30 days.
Vital signs of participants during training | up to 30 days
  The vital signs of participants during training in hospital will be recorded.
Satisfactory assessment | up to 30 days
  Satisfaction of the participants in inspiratory muscle training (IMT) group will be evaluated using a questionnaire at the day of discharged and at 30 days.
Length of stay | up to 120 days
  Length of stay will be assessed by calculating the number of days the patient in the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanhui Liu, MD, PHD, Principal Investigator — Guangdong Provincial People's Hospital, Guangzhou, China.
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Derived] Liu Y, Dai Y, Liu Z, Zhan H, Zhu M, Chen X, Zhang S, Zhang G, Xue L, Duan C, Chen J, Guo L, He P, Tan N. The Safety and Efficacy of Inspiratory Muscle Training for Patients With Acute Myocardial Infarction Undergoing Percutaneous Coronary Intervention: Study Protocol for a Randomized Controlled Trial. Front Cardiovasc Med. 2021 Jan 12;7:598054. doi: 10.3389/fcvm.2020.598054. eCollection 2020. PMID 33511161